CLINICAL TRIAL: NCT01162291
Title: Comparison of Intramuscular Distribution of Different Injection Volumes Via Diffusion Tensor Imaging (DTI)-A Pilot Trial
Brief Title: Comparison of Intramuscular Distribution of Different Injection Volumes Via Diffusion Tensor Imaging (DTI)
Status: Completed | Type: Observational
Sponsor: Kirsten Elwischger (Other)
Responsible Party: Sponsor-Investigator, Kirsten Elwischger, MD, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: MUW-M-MRI01
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: intramuscular; distribution; NaCl; botulinum toxin; muscle; volume; movement; biceps brachii; primary distribution of intramuscular NaCl representative for primary distribution of intramuscular botulinum toxin; shift from extracellular to intracellular viewed by DTI technology; effect of volume; effect of muscle movement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- movement: healthy subjects, randomised to do flexion and extension movements with their left and right elbow joint after intramuscular application of NaCl 2ml in the right musculus biceps brachii, and 1ml in the left musculus biceps brachii
- rest: healthy subjects are randomised to rest after intramuscular application of NaCl 1ml in the left and 2ml in the right musculus biceps brachii

SUMMARY:
The purpose of this experimental pilot study is to assess a positive effect of higher injection volumes of fluid (physiological sodium) in the elbow-flection-muscle (M. biceps brachii) and elbow flexion and extension movements on fluid distribution in the muscle tissue.

DETAILED DESCRIPTION:
Background:

Intramuscular application of Botulinum toxin is used as a successful therapy of many conditions (e.g. spasticity, movement disorders, hypersecretory disorders, ophthalmic disorders, painful conditions, pelvic floor and gastrointestinal disorders, cosmetic applications) Clinical practice shows that even with the use of special guidance techniques (electromyography (EMG), ultrasound, electrical stimulation) to increase accuracy of targeting, botulinum toxin may spread to adjacent sites by diffusion. Different therapy goals request variable diffusion of the toxin, depending on the number of muscles involved and loss of function in the affected area, respectively. There is some evidence that larger injection volume lead to greater distribution and a larger affected area. Thus, animal model showed increased efficacy and decreased systemic side effects of botulinum toxin A in the injected muscle after active or passive manipulation of muscle.

Magnetic resonance imaging (MRI) has the potential to noninvasively probe the amount and motion of intracellular and extracellular water using different sequences. T2-weighted and diffusion tensor sequences are especially useful in the quantification and characterization of the chemical behaviour of water in different (animal) tissue types. To our knowledge there has been no systematically performed in vivo MR study using these imaging techniques in the visualization of intramuscular dilution of fluid in human subjects. However, the in vivo effect on tissue distribution of different injection volumes and active muscle movement in humans via DTI has never been observed.

Hypothesis:

Intramuscular distribution of common saline solutions can be non-invasively quantified by DTI in human subjects. DTI can be used to elucidate if:

* Intramuscular distribution is favoured by larger injection volumes and
* Intramuscular distribution is facilitated by active muscle activity.

Rationale:

The effect of large injection volumes and active muscle activity after injection on intramuscular toxin distribution and uptake remains unclear. Physiological sodium is the carrier material of all preparations of Botulinum toxin, suggesting that physiological sodium or natriumchlorid (NaCl) distribution is representative for toxin primary distribution. Dynamic T2-weighted sequences may monitor the inflow and regional distribution of the infused saline solution.

DTI can non-invasively quantify the amount and directionality of motion of protons in human skeletal muscle and may therefore indirectly allow assumptions on the extra- and intracellular distribution of the infused solution/substance.

Methods:

In this exploratory, investigator blinded pilot study, 10 healthy subjects will be investigated by DTI of the musculi biceps brachii after randomised intramuscular injection of two different injection volumes of NaCl and randomisation to active flexion and extension in the elbow joints versus no active flexion and extension. During each injection dynamic T2 weighted magnetic resonance tomographic sequences will be performed. Subsequently diffusion tensor sequences will be carried out at defined time points.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* willing to participate in this clinical pilot trial
* age 18-80 years old

Exclusion Criteria:

* bleeding disorder or acute bleeding event
* coumarines, warfarin therapy
* any type of medical implant (pacemaker, prosthesis, etc.) not meeting the general safety recommendations for 3 tesla MR imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sycha, Prof., MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Neurology, Vienna, Vienna, Austria

REFERENCES:
- [Background] Hsu TS, Dover JS, Arndt KA. Effect of volume and concentration on the diffusion of botulinum exotoxin A. Arch Dermatol. 2004 Nov;140(11):1351-4. doi: 10.1001/archderm.140.11.1351. PMID 15545544
- [Background] Minamoto VB, Hulst JB, Lim M, Peace WJ, Bremner SN, Ward SR, Lieber RL. Increased efficacy and decreased systemic-effects of botulinum toxin A injection after active or passive muscle manipulation. Dev Med Child Neurol. 2007 Dec;49(12):907-14. doi: 10.1111/j.1469-8749.2007.00907.x. PMID 18039237
- [Background] Kranz G, Haubenberger D, Voller B, Posch M, Schnider P, Auff E, Sycha T. Respective potencies of Botox and Dysport in a human skin model: a randomized, double-blind study. Mov Disord. 2009 Jan 30;24(2):231-6. doi: 10.1002/mds.22336. PMID 18951439
- [Background] Fan RH, Does MD. Compartmental relaxation and diffusion tensor imaging measurements in vivo in lambda-carrageenan-induced edema in rat skeletal muscle. NMR Biomed. 2008 Jul;21(6):566-73. doi: 10.1002/nbm.1226. PMID 18041804
- [Background] Zaraiskaya T, Kumbhare D, Noseworthy MD. Diffusion tensor imaging in evaluation of human skeletal muscle injury. J Magn Reson Imaging. 2006 Aug;24(2):402-8. doi: 10.1002/jmri.20651. PMID 16823776